CLINICAL TRIAL: NCT06752850
Title: A 12-month, Interventional, Open-label, Phase 4 Study in Europe (SHINE) to Investigate the Course of Synovial Hypertrophy as Detected by Joint Ultrasound and MRI in Patients With Haemophilia A on Efanesoctocog Alfa Prophylaxis.
Brief Title: A Study to Investigate the Course of Synovial Hypertrophy in Patients With Haemophilia A on Efanesoctocog Alfa Prophylaxis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.BIVV001-004; 2024-512066-33-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A (Moderate or Severe); Hemophilia, Classic; Haemophilia; Hemophilia; Classic Hemophilia; Synovial Hypertrophy
Keywords: Deficiency, Factor VIII; Factor 8 Deficiency, Congenital; Factor VIII Deficiency; Factor VIII Deficiency, Congenital; Hemophilia A, Congenital; Synovial Membrane; Joint; Prophylaxis
MeSH Terms: conditions — Hemophilia A; Lymphoma, Follicular; Synovitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Treatment Group (Experimental)
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — 50 IU/kg once weekly, Intravenous injection

SUMMARY:
The rationale for conducting this open-label phase 4 study is to assess whether once-weekly prophylaxis with efanesoctocog alfa (50 IU/kg) improves the disease course of existing synovial hypertrophy and prevents the risk of joint bleeds in patients with moderate or severe haemophilia A. The use of imaging assessments will allow for objective detection and monitoring of synovial hypertrophy, and thus expand on the previous findings demonstrating positive effects of once-weekly prophylaxis with efanesoctocog alfa (50 IU/kg) on joint health.

DETAILED DESCRIPTION:
This is a 12-month, multicentre, open-label, non-randomized, interventional single-arm study to assess the course of synovial hypertrophy in previously treated patients ≥12 years of age with moderate or severe haemophilia A achieving high sustained FVIII levels provided by weekly efanesoctocog alfa prophylaxis. To be eligible to enroll in the study, patients must have existing synovial hypertrophy in at least one of the 6 index joints (ankles, elbows, and knees) as assessed by the HEAD-US scoring system. A retrospective data collection on patients' haemophilia, medical, and surgical history will be performed, including a 12-month history of previous treatment and treated bleeding episodes.

The study will start with the Screening Visit, which can be conducted up to 45 days prior to the Baseline Visit (Day 1), to check whether the patient fulfils all the inclusion criteria and none of the exclusion criteria. Patients will have an ultrasound examination of all non-prosthetic index joints at screening. The ultrasound images will be sent for central reading assessment using the HEAD-US scoring system to determine whether the patient has at least one eligible joint required for study inclusion. Once it is confirmed that a patient is eligible for inclusion, he/she will be enrolled in the study and attend a mix of on-site visits and phone call visits. The results from central reading assessment will be sent to the study sites and included in the baseline characteristics of the patients. MRI examinations can be conducted at the Baseline Visit or up to 28 days afterwards. Images from MRI will also be sent for central reading assessment using the International Prophylaxis Study Group (IPSG) MRI scale. The central reading assessment will be sent to the study sites and included in the patient data. Patients will be treated with once-weekly efanesoctocog alfa (50 IU/kg) prophylaxis and will complete the patient diary with their dosing and bleeding information. Assessments will be conducted during the on-site visits, which will occur every 6 months, and during phone call visits, which will occur halfway between these visits. A Safety Follow-up Call will be conducted 14 (+7) days after the End of Treatment (EoT) Visit. Ultrasound and MRI will be used to detect changes in synovial hypertrophy in index joints of patients. The primary endpoint of improvement in existing synovial hypertrophy from baseline to Month 12 as well as the key secondary endpoint of detection of new synovial hypertrophy and change in joint health status from baseline to Month 6 or Month 12 will be assessed using ultrasound and the HEAD-US scoring system.

To obtain 100 eligible index joints, the target is to enroll approximately 35 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol. Parents' or legally designated representatives' consent is required for patients who are <18 years of age or unable to give consent, or as applicable per local laws. Patients who are <18 years of age should provide assent in addition to the parents'/legally designated representatives' consent, if appropriate.
2. Male or female patients who are ≥12 years of age and diagnosed with moderate or severe haemophilia A (defined as ≤5% of normal FVIII clotting activity) at the time of signing the ICF.
3. A female patient is eligible to participate if she is not pregnant at enrolment and does not plan to become pregnant during the study. A woman of child-bearing potential (WOCBP) must have a negative highly sensitive serum pregnancy test at the Screening Visit.
4. Must have received prophylactic treatment per local label with any marketed FVIII product or emicizumab for ≥12 months prior to the Baseline Visit.
5. Have at least one eligible index joint (ankle, elbow, knee).
6. Have 12 months of documented pre-study treatment data on haemophilia prescriptions and on treated bleeding episodes prior to the Baseline Visit.
7. Willingness and the ability of the patient or their legally designated representative to complete training in the use of the study patient diary and to complete the diary throughout the study.

Exclusion Criteria:

1. Blood clotting disorders other than haemophilia A
2. Already on efanesoctocog alfa treatment
3. Positive inhibitor result (assessed by local laboratory) from the Screening Visit, defined as ≥0.6 Bethesda units (BU)/mL.
4. History of inhibitors without successful immune tolerance induction (ITI)

   * Successful ITI is defined as:
   * Negative inhibitor titer (<0.6 BU/mL)
   * FVIII recovery > 66% of expected
   * FVIII half-life ≥ 6 hours
5. ITI performed within the last 2 years prior to the Baseline Visit.
6. Currently receiving treatment with any of the prohibited concomitant medications, as specified by the protocol.
7. Planned major orthopaedic procedure in any eligible index joint during the course of the study.
8. Patients are not eligible for participation in the study if they cannot undergo MRI assessments at the Baseline Visit.
9. Patients with known hypersensitivity to the active substance or to any of the excipients.
10. Patient not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or patients potentially at risk of noncompliance to study procedures.
11. Enrolment in a concurrent clinical interventional study, or intake of an investigational medicinal product (IMP), within 3 months prior to inclusion in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) synovial hypertrophy domain score decrease. | Baseline to 12 months
  At least 1 point decrease in HEAD-US synovial hypertrophy domain score at Month 12 (for joints with a domain score of 1 or 2 at baseline).

SECONDARY OUTCOMES:
Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) synovial hypertrophy domain score increase. | Baseline to 6 or 12 months
  At least 1 point increase in HEAD-US synovial hypertrophy domain score at Month 6 or Month 12 for joints with no synovial hypertrophy at baseline (domain score of 0).
International Prophylaxis Study Group (IPSG) magnetic resonance imaging (MRI) | Baseline to 12 months
  Change from baseline in total/domain scores of International Prophylaxis Study Group (IPSG) MRI per patient and per joint at Month 12.
Haemophilia Joint Health Score (HJHS) | Baseline to 12 months
  Change from baseline in total/domain scores of HJHS per patient and per joint at Month 12.
Patient Reported Outcome (PRO) of Pain Intensity | Baseline to 6 month and 12 months
  Use of PROMIS SF v2.0 to measure change in patient-reported pain intensity from baseline.
Patient Reported Outcome of Pain Interference | Baseline to 6 month and 12 months
  Use of PROMIS SF v2.0 to measure change in patient-reported pain interference from baseline.
Patient Reported Outcome of Physical Function | Baseline to 6 month and 12 months
  Use of PROMIS SF v2.0 to measure change in patient-reported physical function from baseline.
Patient Reported Outcome of 5-level EuroQol-5 dimensions [EQ-5D-5L] score | Baseline to 6 month and 12 months
  Changes from baseline of patient self-care, usual activities, pain/discomfort, anxiety/depression.
Hemo-FAST scoring | Baseline to 12 months
  Assess functional mobility in PWH. The Hemo-Fast tool is comprised of the Patient-reported outcome part and a Clinician-reported outcome (ClinRO) part, with a score of 0 to 100, with zero being the best possible joint health status. The change from baseline to month 12 will be evaluated.
Change in annualized bleeding rate (ABR) and annualized joint bleeding rate (AjBR) (spontaneous, traumatic). | 12 months prior to on-study period (retrospective) to 12 months after start of study intervention (prospective)
The occurrence of treatment-emergent adverse events (TEAEs) leading to treatment discontinuation, serious TEAEs, and adverse events of special interest (AESIs). | 12 months, +14 (+7days) after the last IMP dose
Patient-Reported Treatment Preference Questionnaire | 12 month
  A 2-item treatment survey developed to evaluate perceived impact of treatment.
Qualitative Exit Interview | Within 14 days after EoT Visit
  60-minute Telephone Interview patient reported preference for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Sobi AB
Locations (10):
- Italy (3):
  - Sobi Investigational Site, Milan
  - Sobi Investigational Site, Naples
  - Sobi Investigational Site, Rozzano
- Sobi Investigational Site, Oslo, Norway
- Spain (4):
  - Sobi Investigational Site, Barcelona
  - Sobi Investigational Site, Madrid
  - Sobi Investigational Site, Seville
  - Sobi Investigational Site, Valencia
- Sweden (2):
  - Sobi Investigational Site, Gothenburg
  - Sobi Investigational Site, Malmo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents. Patient level data will be anonymized and study documents, if applicable will be redacted to protect the privacy of trial participants.
URL: http://www.sobi.com/en/policies